CLINICAL TRIAL: NCT02474810
Title: Comparison of an Intensive Versus a Standard Hemodialysis Central Venous Catheter Dysfunction Protocol Using Alteplase
Brief Title: Intensive Versus Standard Hemodialysis CVC Dysfunction Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Dialysis Catheter Protcols
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Chronic Renal Insufficiency
Keywords: central venous catheters; hemodialysis; thrombosis; tissue plasminogen activator
MeSH Terms: conditions — Renal Insufficiency, Chronic; Thrombosis | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive (Experimental): In the Intensive Protocol, alteplase intervention is administered to all catheters based on blood flow and/or line reversal
  Interventions: Drug: Alteplase
- Standard (Experimental): In the Standard Protocol, alteplase intervention is administered to all catheters based only on blood flow.
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Alteplase — Alteplase for CVC dysfunction.
  Other Names: Cathflo; rt-PA

SUMMARY:
Central venous catheters (CVCs) are used for vascular access by approximately 56% of our 380 hemodialysis (HD) patients at the Capital Health Renal Program. The major complication of these catheters includes thrombosis and infection. Catheter locking solutions such as recombinant tissue plasminogen activator (rt-PA), Alteplase (Cathflo®) are used to treat and prevent clotting of the catheter during HD treatments and during the interdialytic period. Evidence to guide the use of rt-PA is limited. This quality assurance project will compare the effectiveness and cost of an intensive versus a standard catheter dysfunction protocol for rt-PA in HD patients.

DETAILED DESCRIPTION:
The proposed study will be a retrospective cohort study of consecutive HD patients conducted at a HD unit using two catheter dysfunction protocols during January 2013 to Septebmer 2013. In the Intensive Protocol, rt-PA intervention is administered to all catheters based on blood flow and/or line reversal. In the Standard Protocol, rt-PA intervention is administered to all catheters based only on blood flow.

ELIGIBILITY:
Inclusion Criteria:

* All adults undergoing HD with a tunneled CVC (both newly inserted CVCs as well as pre-existing CVCs) will be included.

Exclusion Criteria:

* Patients were excluded from using the CVC dysfunction protocols if they had a known allergy or intolerance to rt-PA.
* A physician order to proceed with the CVC dysfunction protocols was required if they met one of the following criteria:
* CVC line insertion or exchange within 72 hours;
* any surgery, organ biopsy, obstetrical delivery within 72 hours;
* active bleeding; bleeding disorders; hemoglobin decrease greater than 20 g/L over 2 weeks;
* active pericarditis; arterial puncture within 48 hours;
* bacteremia with positive blood cultures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Alteplase use | 9 months
  Incident rate of rt-PA uses includes the numerator which will consist of the number of HD sessions during which a patient was administered rt-PA for catheter malfunction and the denominator will be the time period at risk in catheter days.

SECONDARY OUTCOMES:
Rate of bacteremia | 9 months
  Rate of bacteremia will include the numberator which will consit of the number of definite or probable catheter related bacteremia events and the decominator will be the time period at risk in catheter days.
Cost of alteplase | 9 months
  Cost of rt-PA will be calculated per TLD for the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jo-Anne S Wilson, PharmD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Capital Health District Authority, Department of Medicine, Division of Nephrology, Halifax, Nova Scotia, Canada